CLINICAL TRIAL: NCT02906176
Title: A Clinical Trail to Investigate the Influence of SLCO2B1 Polymorphism on the Pharmacokinetic Characteristics of Voriconazole in CYP2C19 Poor Metabolizers
Brief Title: Influence of SLCO2B1 Polymorphism on the PK of Voriconazole in CYP2C19 PM
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, SeungHwan Lee, Assistant Professor, Seoul National University Hospital
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: CYP2C19-SLCO2B1
Record Dates: First submitted 2016-09-12; First posted 2016-09-19 (Estimated); Last update posted 2017-10-25 (Actual); Status verified 2016-09

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Voriconazole; Infusions, Intravenous; Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- SLCO2B1 wild type (Experimental): Vfend (voriconazole) 200 mg intravenous infusion during 1.5 h (Day 1) - washout period - Vfend (voriconazole) 200 mg tablet once (Day 8)
  Interventions: Drug: Vfend (voriconazole) intravenous infusion; Drug: Vfend (voriconazole) tablet
- SLCO2B1 variant (Experimental): Vfend (voriconazole) 200 mg intravenous infusion during 1.5 h (Day 1) - washout period - Vfend (voriconazole) 200 mg tablet once (Day 8)
  Interventions: Drug: Vfend (voriconazole) intravenous infusion; Drug: Vfend (voriconazole) tablet

INTERVENTIONS:
Drug: Vfend (voriconazole) intravenous infusion — Vfend (voriconazole) 200 mg intravenous infusion during 1.5 h
  Other Names: IV
Drug: Vfend (voriconazole) tablet — Vfend (voriconazole) 200 mg tablet once
  Other Names: Oral

SUMMARY:
A clinical trail to investigate the influence of SLCO2B1 polymorphism on the pharmacokinetic characteristics of voriconazole in CYP2C19 poor metabolizers

ELIGIBILITY:
Inclusion Criteria:

* Healthy male volunteer who is a CYP2C19 Poor metabolizer with rs3781727 SNP wild or variant genotype

Exclusion Criteria:

* History of clinically significant respiratory, cardiovascular, renal, hepatic, hematologic, neurological disorder

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2016-09; Primary Completion 2016-11 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic outcome - Maximum plasma concentration (Cmax) | predose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72 hours post-dose
Pharmacokinetic outcome - Area under the plasma concentration versus time curve (AUC) | predose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72 hours post-dose

CONTACTS AND LOCATIONS:
Overall Officials: SeungHwan Lee, MD., PhD., Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital Clinical Trial Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided